CLINICAL TRIAL: NCT06739733
Title: Effectiveness of Soft Robotic Glove Versus EMS on Hand Function and Quality of Life in Stroke Survivors. A Randomized Clinical Trial
Brief Title: Effectiveness of Soft Robotic Glove Versus EMS on Hand Function and Quality of Life in Stroke Survivors (RCT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/748
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SRG (Experimental)
  Interventions: Diagnostic Test: SRG
- EMS (Active Comparator)
  Interventions: Diagnostic Test: EMS

INTERVENTIONS:
Diagnostic Test: SRG — Soft robotic gloves stimulation 30-minute sessions, 5 times per week upto 8 week Soft robotic gloves are assistive devices designed to enhance hand function for individuals with disabilities or injuries. These gloves use flexible materials, such as silicone or fabric, combined with pneumatic or cable-driven mechanisms to mimic natural hand movements. They provide assistance for gripping, holding, or manipulating objects, often controlled by sensors or user inputs. Soft robotic gloves are lightweight, adaptable, and offer rehabilitation potential, helping restore motor function in conditions like stroke or spinal cord injury. They are increasingly used in clinical and home-based therapy settings.
  Arms: SRG
Diagnostic Test: EMS — Electrical muscle stimulation 30-minute sessions, 5 times per week upto 8 weeks.
  Electrical Muscle Stimulation (EMS) is a technique that uses electrical impulses to contract muscles, often used for rehabilitation, strength training, or pain management. Electrodes placed on the skin deliver controlled currents to target specific muscle groups, mimicking natural nerve signals. EMS is commonly used in physiotherapy to prevent muscle atrophy, improve circulation, and enhance recovery after injury. It is also utilized in fitness and sports for performance enhancement. Safe and non-invasive, EMS can be adjusted for therapeutic or functional goals.
  Arms: EMS

SUMMARY:
This study will evaluate the effectiveness of soft robotic gloves versus electrical muscle stimulation (EMS) in improving hand function and quality of life in stroke survivors. Stroke often leads to impaired hand mobility, impacting daily activities and reducing overall quality of life. Soft robotic gloves, designed to assist with hand movement, will provide mechanical support and encourage voluntary muscle activity. EMS, on the other hand, will stimulate muscle contraction through electrical impulses, potentially enhancing muscle strength and coordination.

DETAILED DESCRIPTION:
Participants will be divided into two groups: one will receive treatment using soft robotic gloves, and the other with EMS. Outcomes will be assessed using standardized hand function tests and quality-of-life questionnaires over a specified period. Results are expected to indicate that both interventions will improve hand function and quality of life, with the robotic gloves showing a marginally greater improvement in dexterity and grip strength, while EMS will yield benefits in muscle reactivation and endurance. Stroke survivors in the robotic glove group are anticipated to report greater ease in performing daily tasks, while the EMS group will note an increase in muscle engagement.

ELIGIBILITY:
Inclusion Criteria:

* Had ischemic or hemorrhagic stroke ≤6 months.
* Mini-mental status exam scores > 24(7).
* GCS score 11 to 15(2)
* FMA-UE score < 21(3)

Exclusion Criteria:

* Participants with severe vision or hearing impairment.
* Neurological disorders including epilepsy, Alzheimer's disease, vertigo, Parkinson disease, and , muscular disorders which limit functional activity (OA, RA, etc).
* Peripheral vestibular disorder.
* Medications that affect balance, severe cardiovascular conditions, recent lower limb injury or surgery.
* Contraindications for EMS: Patients with certain medical conditions, such as pacemakers, implantable cardioverter-defibrillators, or metal fragments in their body, that contraindicated the use of EMS were excluded.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The Fugl-Meyer Upper Extremity Assessment (FMA-UE) | 12 Months
  The Fugl-Meyer Upper Extremity Assessment (FMA-UE) is a standardized tool used to evaluate motor function, sensation, coordination, and joint motion in individuals with upper limb impairments, often post-stroke. It is based on a hierarchical framework of motor recovery, covering movements from basic reflexes to voluntary motor control. The assessment includes various sections focusing on shoulder, elbow, forearm, wrist, hand, and coordination. Each item measures specific movement tasks, allowing therapists to track progress over time. The FMA-UE is widely used in clinical settings for its reliability and validity in evaluating upper extremity function.
  Scoring
  The FMA-UE has 33 items, each scored on a 3-point scale:
  0 = Cannot perform
  1. = Partially performs
  2. = Fully performs
  The total score ranges from 0 to 66 points (higher scores indicate better motor function).
The Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) | 12 months
  The Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) is a shortened version of the DASH outcome measure used to assess physical function and symptoms in individuals with upper extremity conditions. It consists of 11 questions evaluating difficulty in performing daily activities, severity of symptoms (pain, tingling, weakness), and social and emotional impacts. The QuickDASH is designed for fast administration and is applicable across various musculoskeletal disorders. It provides insight into functional limitations, helping guide treatment planning.
  Scoring
  Each item is rated on a 1-5 Likert scale (1 = no difficulty, 5 = extreme difficulty).
  Scores are averaged, transformed into a scale of 0 to 100 (0 = no disability, 100 = most severe disability).
  An optional Work and Sports/Performing Arts module adds context-specific insights.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad block garden town canal road, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No